CLINICAL TRIAL: NCT05920811
Title: Patient Satisfaction With Conventional Maxillary Obturator Versus Fully Digital Fabricated With 3D Printing: a Randomized Crossover Trial
Brief Title: Patient Satisfaction for Digital Versus Conventional Maxillary Obturator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Mohammed Amer, lecturer, Tanta University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: prosth 6/23
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Maxillofacial Prosthesis User
Keywords: maxillary obturator, selective laser melting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- conventional obturator (Active Comparator): maxillary obturator fabricated from cast metal framework, heat-cured acrylic resin
  Interventions: Other: conventional obturator
- 3 d printed obturator (Experimental): 3d printed obturator with full digital workflow ( intraoral scanning, made of selective laser melting, 3d printed resin
  Interventions: Other: 3 d printed obturator

INTERVENTIONS:
Other: conventional obturator — restoration of midline maxillary defect with obturator made of cast metal , heat cure acrylic resin
  Arms: conventional obturator
Other: 3 d printed obturator — restoration of midline maxillary defect with obturator made of SLM metal , 3 d printed resin
  Arms: 3 d printed obturator

SUMMARY:
Evidence regarding the performance of digital obturators totally fabricated using 3D printing is insufficient. This prospective randomized crossover study aimed to evaluate patient satisfaction with conventional maxillary obturator and totally full digitally fabricated obturator. Patient satisfaction was evaluated using two scales: The Obturator Functioning Scale" and "The Patient and operator-centered outcomes were assessed through two visual analog scale (VAS) questionnaires.

DETAILED DESCRIPTION:
The use of digital technologies in the fabrication of maxillofacial prostheses has been described. Additive manufacturing offers a more convenient and more efficient process with reduced material waste compared with traditional subtractive technique. Although Prosthetic rehabilitation with Conventional maxillary obturator prosthesis fabricated with a casted metal framework using, heat-cured acrylic resin can restore oral function and facial esthetics following maxillectomy. But it is time-consuming and labor-intensive. Multiple sources of errors can accumulate during the laboratory steps, resulting in a misfit of the framework. In this study All patients received a conventional obturator for 6 months, after a washout period of one week, they use the digital one. The Obturator Functioning Scale" and "The Patient and operator-centered outcomes were assessed through two visual analog scale (VAS) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patients with hemimaxillectomy defect (Aramany class 1)
* almost edentulous mandible with healthy remaining teeth,
* mouth opening is not less than 25 mm, intact soft palate
* participants were not exposed to radiotherapy or chemotherapy in the previous year

Exclusion Criteria:

* patients with physical or mental disorders.
* patients still receiving radio or chemotherapy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
obturator functioning scale | 6 months
  The Obturator Functioning Scale ( minimum value is "1"and maximum value is "5"
patient outcome the treatment time, on the self-perception of the applied impression protocol in terms of general convenience, anxiety, taste, nausea sensation and possible pain sensation. | 6 months
  questions focused on general convenience, anxiety, taste, nausea sensation and possible pain sensation, assessed through visual analogue scale (VAS)
operator outcome | 6 months
  Questions focused on the treatment time, on the self-perception of the applied impression

CONTACTS AND LOCATIONS:
Overall Officials: marwa M Amer, Principal Investigator — Tanta University
Locations (1):
- marwa Mohammed Amer, Tanta, ElGharbia, Egypt